CLINICAL TRIAL: NCT06957938
Title: A Prospective, Multi-centered, Randomized Phase III Study to Compare Neoadjuvant Chemotherapy Combined With PD-1 Inhibitor Versus Neoadjuvant Chemotherapy in Locally Advanced Laryngeal and Hypopharyngeal Carcinoma
Brief Title: Comparing Neoadjuvant Chemotherapy Combined With PD-1 Inhibitor Versus Neoadjuvant Chemotherapy in Locally Advanced Laryngeal and Hypopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Sun Yat-sen University Cancer Center (SUSUCC) (Unknown); Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yu Wang, M.D., Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRECEDE; 2504318-4 (Other: Fudan University Shanghai Cancer Center)
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Laryngeal Carcinoma; Hypopharyngeal Carcinoma
Keywords: Neoadjuvant chemotherapy; Induction chemotherapy; Immunotherapy; anti-PD-1 antibody; PD-1 inhibitor; Tislelizumab; surgery; radiation; Locally advanced disease; Laryngeal preservation; Laryngeal cancer; Hypopharyngeal cancer; Head and neck cancer; Head and neck squamous cell carcinoma
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Neoadjuvant Therapy; Surgical Procedures, Operative; Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant chemotherapy combined with Tislelizumab (Experimental): Neoadjuvant chemotherapy combined with Tislelizumab, followed by chemo-radiation or surgery and adjuvant (chemo-)radiation, then maintenance therapy of Tislelizumab.
  Interventions: Drug: Neoadjuvant Chemotherapy (NACT); Drug: Neoadjuvant and maintenance Tislelizumab; Radiation: Concurrent chemo-radiotherapy (CCRT); Procedure: Surgery and adjuvant (chemo-)radiotherapy
- Neoadjuvant chemotherapy (Active Comparator): Neoadjuvant chemotherapy, followed by chemo-radiation or surgery and adjuvant (chemo-)radiation.
  Interventions: Drug: Neoadjuvant Chemotherapy (NACT); Radiation: Concurrent chemo-radiotherapy (CCRT); Procedure: Surgery and adjuvant (chemo-)radiotherapy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy (NACT) — Neoadjuvant Chemotherapy with paclitaxel (or albumin - bound paclitaxel) and cisplatin
Drug: Neoadjuvant and maintenance Tislelizumab — Neoadjuvant and maintenance Tislelizumab
  Arms: Neoadjuvant chemotherapy combined with Tislelizumab
Radiation: Concurrent chemo-radiotherapy (CCRT) — Concurrent chemo-radiotherapy (CCRT), with cisplatin-based chemotherapy
Procedure: Surgery and adjuvant (chemo-)radiotherapy — Definitive surgery, with adjuvant (chemo-)radiotherapy, depending on pathologic findings.

SUMMARY:
Neoadjuvant chemotherapy combined with immunotherapy has achieved promising pathological remission rates in locally advanced head and neck squamous cell carcinoma and has offered new hope for patients with locally advanced laryngeal and hypopharyngeal cancer. In our center's previous phase II study on locally advanced laryngeal and hypopharyngeal cancer, neoadjuvant chemotherapy combined with immunotherapy showed good 1 - year laryngeal preservation rate and 1 - year PFS rate. However, in locally advanced laryngeal and hypopharyngeal cancer, whether neoadjuvant chemotherapy combined with PD-1 inhibitor, compared with neoadjuvant chemotherapy, can improve laryngeal preservation survival, event - free survival and overall survival remains unclear.

Thus, this study aims to explore in locally advanced laryngeal and hypopharyngeal cancer whether neoadjuvant immuno - chemotherapy, compared with neoadjuvant chemotherapy, can improve laryngeal preservation survival and bring benefits in quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have signed the informed consent form and are willing to complete the study according to the protocol.
2. Age ≥18 years and ≤75 years.
3. Histologically confirmed squamous cell carcinoma of the larynx or hypopharynx.
4. Locally advanced laryngeal or hypopharyngeal cancer that requires total laryngectomy and is amenable to total laryngectomy according to surgical assessment.
5. At least one measurable lesion before treatment, which meets the criteria for "measurable lesion" according to RECIST 1.1 criteria.
6. An expected survival of >3 months.
7. ECOG performance status of 0-1.
8. Adequate organ function, meeting the following requirements:

   1. Absolute neutrophil count (ANC) ≥1.5×10^9/L;
   2. Platelet count ≥100×10^9/L;
   3. Hemoglobin ≥9 g/dL;
   4. Serum albumin ≥2.8 g/dL;
   5. Total bilirubin ≤1.5×ULN, ALT, AST, and/or ALP ≤3×ULN;
   6. Serum creatinine ≤1.5×ULN and creatinine clearance ≥60 mL/min (Cockcroft-Gault, see Appendix III);
   7. Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤1.5×ULN (patients on stable doses of anticoagulant therapy, such as low-molecular-weight heparin or warfarin, with INR within the therapeutic range of the anticoagulant, are eligible).
9. Patients with hepatitis B virus (HBV) infection, as well as inactive/asymptomatic HBV carriers, or those with chronic or active HBV, will be allowed to enroll if HBV DNA <500 IU/mL (or 2500 copies/mL) at screening. Patients who are positive for hepatitis C antibody will be allowed to enroll if HCV-RNA is negative at screening.
10. Women of childbearing potential must have a negative urine or serum pregnancy test within ≤7 days before treatment. They must also agree to use an accepted method of contraception (e.g., intrauterine device, oral contraceptives, or condoms) during the study treatment period, as well as for at least 3 months after the last dose of PD-1 inhibitor and at least 6 months after the last dose of chemotherapy.
11. Male subjects who have not been sterilized must agree to use an accepted method of contraception (e.g., intrauterine device, oral contraceptives, or condoms) during the study treatment period, as well as for at least 3 months after the last dose of PD-1 inhibitor and at least 6 months after the last dose of chemotherapy.

Exclusion Criteria:

1. Patients who have been confirmed to have distant metastasis on imaging assessment before treatment.
2. Patients who have previously received immune checkpoint inhibitor therapy.
3. Patients who have previously received radiotherapy to the head and neck region.
4. Patients who have had or currently have other malignancies (except for malignancies that have been cured and have been cancer-free for more than 5 years, such as basal cell carcinoma of the skin, cervical carcinoma in situ, and papillary thyroid cancer); if a patient has both hypopharyngeal cancer and esophageal cancer, and the esophageal lesion and hypopharyngeal lesion are anatomically non-adjacent, they should be diagnosed with multiple primary tumors and will not be eligible for enrollment.
5. Uncontrolled cardiac symptoms or diseases, such as: a. NYHA Class II or higher heart failure; b. unstable angina; c. myocardial infarction within the past year; d. clinically significant supraventricular or ventricular arrhythmias that are not well controlled with medication.
6. Patients who have received any of the following treatments:

   1. Received any investigational drug within 4 weeks before the first dose of the study drug.
   2. Enrolled in another clinical study concurrently, unless it is an observational (non-interventional) clinical study.
   3. Require systemic treatment with corticosteroids (more than 10 mg prednisone equivalent per day) or other immunosuppressive agents within 2 weeks before the first dose of the study drug, except for corticosteroids used for local inflammation and prevention of allergies and nausea/vomiting. Other special circumstances should be discussed with the investigator. In the absence of active autoimmune disease, the use of inhaled or topical steroids and adrenal corticosteroid replacement at doses greater than 10 mg/day prednisone equivalent is permitted.
   4. Received anti-tumor vaccines or live vaccines within 4 weeks before the first dose of the study drug (if the patient has received a COVID-19 vaccine, the interval between vaccination and treatment should be more than 2 weeks).
   5. Underwent major surgery or had a severe injury within 4 weeks before the first dose of the study drug.
7. Patients who have had a severe infection (CTCAE > Grade 2) within 4 weeks before the first dose of the study drug, such as severe pneumonia, bacteremia, or infectious complications requiring hospitalization; baseline chest imaging showing active pulmonary inflammation; symptoms and signs of infection within 4 weeks before the first dose of the study drug or requiring oral or intravenous antibiotic treatment.
8. Patients with active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); however, this does not include autoimmune hypothyroidism treated with a stable dose of thyroid hormone replacement therapy; type 1 diabetes treated with a stable dose of insulin; vitiligo or childhood asthma/allergies that have healed and do not require any intervention in adulthood.
9. Patients with a history of immunodeficiency, including positive HIV test results, or those with other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation.
10. Patients with a history of interstitial lung disease (excluding radiation pneumonitis that has not been treated with corticosteroids) or non-infectious pneumonia.
11. Patients with active tuberculosis infection identified through history or CT scan, or those with a history of active tuberculosis infection within 1 year before enrollment, or those with a history of active tuberculosis infection more than 1 year ago that was not properly treated.
12. Patients with active hepatitis B (HBV DNA ≥500 IU/mL or 2500 copies/mL) or hepatitis C (positive hepatitis C antibody and HCV-RNA above the lower limit of detection of the assay).
13. Patients with a known history of abuse of psychoactive drugs, alcoholism, or drug addiction.
14. Pregnant or breastfeeding women.
15. Patients who, in the investigator's judgment, have other factors that may force them to discontinue the study prematurely, such as having other serious diseases (including mental illnesses) requiring concurrent treatment, severely abnormal laboratory values, family or social factors, or conditions that may affect the patient's safety or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
2-year Laryngectomy-free Survival Rate | 2 year
  Laryngectomy-free survival (LFS) is defined as the time from randomization to the first occurrence of local recurrence, total laryngectomy, or death, with the time calculated based on the first event that occurs.

SECONDARY OUTCOMES:
Early response rate | day 14 to day 21
  Early response rate is defined as the proportion of patients achieving a complete response [CR] or partial response [PR] in the primary tumor after one cycle of neoadjuvant therapy
Objective response rate to neoadjuvant therapy | day 56 to day 63
  Objective response rate to neoadjuvant therapy is defined as the proportion of patients achieving a complete response (CR) or partial response (PR) in the primary tumor and cervical lymph nodes after three cycles of neoadjuvant therapy.
2-year Event-free Survival Rate | 2 year
  Event-free survival (EFS), defined as the time from randomization to the first occurrence of any of the following events: disease progression precluding surgical treatment, local recurrence, distant metastasis, or death from any cause, whichever occurs first.
2-year Overall Survival Rate | 2 year
  Overall Survival (OS), defined as the time from randomization to death from any cause.
2-year Laryngectomy-free Survival Rate with a functional larynx | 2 year
  Laryngectomy-free survival with a functional larynx (fLFS), defined as the time from randomization to the occurrence of an endpoint event, which includes: evidence of local recurrence; total laryngectomy; death; or survival at 2 years with tracheostomy, nasogastric tube, or gastrostomy.
2-year Local Recurrence-Free Survival Rate | 2 year
  Local Recurrence-Free Survival (LRFS): Defined as the time from randomization to the first documentation of local recurrence or to death from any cause.
2-year Distant Metastasis-Free Survival Rate | 2 year
  Distant Metastasis-Free Survival (DMFS): Defined as the time from randomization to the first documentation of distant metastasis or to death from any cause, whichever occurs first.
Adverse event | 2 year
  Adverse events, defined as any untoward medical occurrence in a clinical trial subject after randomization up to 2 years post-randomization, which does not necessarily have a causal relationship with the treatment.
Quality of life | 2 year
  Quality of life, assessed based on disease-related symptoms and quality of life using the EORTC Quality of Life Questionnaire Head and Neck (H&N)-35 score. For scores related to speech and swallowing function, the higher score indicates more severe symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Wang, M.D., professor, Chief, Principal Investigator — Department of head and neck surgery, Fudan University Shanghai Cancer Center
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fang Q, Xu P, Cao F, Wu D, Liu X. PD-1 Inhibitors combined with paclitaxel (Albumin-bound) and cisplatin for larynx preservation in locally advanced laryngeal and hypopharyngeal squamous cell carcinoma: a retrospective study. Cancer Immunol Immunother. 2023 Dec;72(12):4161-4168. doi: 10.1007/s00262-023-03550-z. Epub 2023 Oct 7. PMID 37804437
- [Background] Ou X, Zhai R, Wei W, Chen J, Ou D, Liao T, Xu T, Zhu Y, Wang Y, Huang S, Shi R, Wu B, Chen T, Li Y, Yang Z, Zhou C, Liu Y, Jiang Z, Zeng M, Liu X, Ji D, Ying H, Zhang Z, Hu C, Lu X, Ji Q, He X, Wang Y. Induction Toripalimab and Chemotherapy for Organ Preservation in Locally Advanced Laryngeal and Hypopharyngeal Cancer: A Single-Arm Phase II Clinical Trial. Clin Cancer Res. 2024 Jan 17;30(2):344-355. doi: 10.1158/1078-0432.CCR-23-2398. PMID 37955629